CLINICAL TRIAL: NCT03671486
Title: Observational Study to Investigate the Probability of Colonization with Group B Streptococcus (GBS) of Pregnant Women Who Were Negative for GBS in the First Trimester of Pregnancy
Brief Title: Colonization with Group B Streptococcus During Pregnancy
Acronym: PROBIGEST
Status: Completed | Type: Observational
Sponsor: ProbiSearch SL (Industry)
Collaborators: Casen Recordati S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: STB/17.02.1
Record Dates: First submitted 2018-08-30; First posted 2018-09-14 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2020-10

CONDITIONS: Gestational Mother; Streptococcus Agalactiae Infection
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Vagino-rectal exudate from participant will be collected at visit 1 and 3 to detect the presence of Group B Streptococcus. After that, they will be destroyed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- GBS-negative pregnant women: One Hundred Healthy GBS-negative pregnant women will be follow-up since the first trimester of pregnancy until one month post-delivery

SUMMARY:
An observational study to estimate the probability of pregnant women, who were GBS-negative in the first trimester of pregnancy become GBS-positive at the end of pregnancy. It is an observational. One hundred pregnant women in the first trimester of pregnancy (11 ± 2 weeks) will be invite to participate in this prospective study. If accept, a vagino-rectal swab will collected for a GBS detection analysis. When negative, participants will be follow by their gynecologist with the normal routine procedures. During 35 week of pregnancy a vagino-rectal swab will be collected and analyzed to detect GBS. Then, a final visit will be completed one month after delivery.

DETAILED DESCRIPTION:
Healthy pregnant women reporting to the clinic in their first trimester of pregnancy (week 11 ± 2 weeks of pregnancy) will be asked to participate in this study. Participation will be voluntary and written informed consent will be obtained from each participant. The study visits will take place in the hospital.

At Visit 1, the inclusion and exclusion criteria will be verified. After signing the informed consent, a physical examination will be performed in addition to a vaginal-rectal swab to detect if they are GBS-negative. Information on the demographic profile and medical history will be collected. The investigator will explain to the participant that she cannot use any probiotic during the course of the study.

At Visit 2, within 21-23 weeks ± 4 days of gestation, the inclusion and exclusion criteria will be reviewed. If the result of the microbiological analysis of the vaginal-rectal exudate is negative, the pregnant women shall continue in the study. A physical examination will be performed. Adverse Events occurring from the time of study inclusion will be recorded.

At the third visit (Visit 3, 35 weeks ± 4 days of gestation), all participants continuing in the study will undergo a general physical examination. A sample of vagino-rectal exudate will be collected. Adverse Events occurring during the period between Visit 2 and Visit 3 will be recorded.

During Visit 4 (1 month after delivery), all participants will have a general physical examination. Adverse Events occurring since Visit 3 will be recorded. Data will be collected on the delivery and occurrence of early- or late-onset GBS sepsis in the newborn during the first month of life.

ELIGIBILITY:
Inclusion Criteria:

Healthy pregnant women, adults (≥ 18 years and under 45 years). Before/during week 13 of gestation. Signing of informed consent.

Exclusion Criteria:

Multiple pregnancy.

Fetal complications.

History of premature delivery/miscarriage in the second trimester. Significant maternal medical complications.

HIV-positive.

Women who are immunocompromised (for example, patients with cancer and transplant who are taking certain immunosuppressive drugs, patients with hereditary diseases that affect or could affect the immune system).

History of significant gastrointestinal disease (e.g., prior gastrointestinal resection, current diarrhea, inflammatory bowel disease).

Heart failure and cardiac medical history (e.g. artificial heart valve, medical history of infective endocarditis, rheumatic fever or cardiac malformation).

Use of other probiotics during the current pregnancy.

Uncertainty of the investigator regarding the willingness or capacity of the participant to comply with the requirements of the protocol.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women
Study Population: 100 pregnant women GBS (-)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Participants (%) with a vaginal-rectal detection of Group B Streptococcus. | 6 months
  Percentage of participants with a vaginal-rectal detection of Group B Streptococcus at the end of the study.

SECONDARY OUTCOMES:
Composition of the microbiota of vaginal-rectal exudates | 6 months
  Amounts (log(CFU/mL) and identification of bacterial species detected by culture in vaginal-rectal exudates from pregnant women
Premature membrane rupture | 7 months
  % of participants with premature rupture of the membranes
Premature detachment of the placenta | 7 months
  % of participants with premature detachment of the placenta
Premature delivery | 7 months
  % of participants with premature delivery
Pregnancy complications | 7 months
  % of participants with pregnacy complications
Newborns with early onset sepsis | 7 months
  Percentage of newborns with early onset sepsis
Newborns with late onset sepsis | 7 months
  Percentage of newborns with late onset sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Susana Manzano, PhD, Study Chair — ProbiSearch SL
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided